CLINICAL TRIAL: NCT01885754
Title: Characterization of Peripheral Muscle Function in Patients With Non-small-cell Lung Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Didier Saey, PhD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Other Study IDs: 20878
Record Dates: First submitted 2013-02-13; First posted 2013-06-25 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Non-Small-cell Lung Cancer
Keywords: Biopsy; Maximal incremental cardiopulmonary test; Muscle strength test; magnetic stimulation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Quadriceps Biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lung cancer patient with cachexia: Muscle lumbar area < 55cm2/m2 for men and < 39 cm2/m2 for women
- Lung cancer patients without cachexia: Muscle lumbar area over 55cm2/m2 for men and 39 cm2/m2 for women

SUMMARY:
Rationale: With 1.6 million new cases diagnosed each year and 1.3 million deaths, lung cancer is the leading cancer-related death worldwide and it represents a pressing health issue. Patients with lung cancer are more likely to experience cachexia, a severe debilitating disorder causing fatigue, weight loss, muscle wasting and associated with reduced physical function, increased chemotherapy toxicity and reduced survival. This syndrome occurring in about 80% of advanced cancer patients is the direct cause of death in about 20% of cases. However, despite the importance of cachexia in lung cancer, its mechanisms ans its relation with muscle function and effort tolerance are still unknown.

Aim: To explore muscle function, signaling pathways and its relationship to impaired functional capacity of patients with non-small-cell lung cancer(NSCLC); depending of whether they have cachexic state at diagnosis.

Methods: This study will be conducted at the Institut universitaire de cardiologie et de pneumologie de Québec. 56 patients newly diagnosed of NSCLC will be recruited and separated whether or not they have a cachexic state. The evaluation will need two visits separated by 5 days.

During the evaluation the following tests will be done:

* Anthropometric measures
* Level of daily physical activity
* Pulmonary function test
* Maximal incremental cardiopulmonary exercise test on ergocycle
* Endurance test on ergocycle
* Muscle function tests
* Magnetic stimulation
* Quadriceps biopsy

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a primary lung cancer diagnosis

Exclusion Criteria:

* Already have undertaken surgery, chemotherapy or radiotherapy treatment
* Having an other cancer in the last five years
* Taking anticoagulation therapy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Maximal quadriceps strength | 1 day (at the time of the diagnosis before any treatment)

SECONDARY OUTCOMES:
Exercise capacity | 1 day (at the time of the diagnosis before any treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Saey, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada